CLINICAL TRIAL: NCT01728142
Title: Comparison of the Defense Automated Neurobehavioral Assessment (DANA) Brief Exam to the Automated Neuropsychological Assessment Metrics (ANAM) Battery in the Evaluation of Cognitive Changes During Concussion Recovery
Brief Title: Comparison of the DANA to the ANAM in the Evaluation of Cognitive Changes After Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, jack tsao, Director, TBI Programs, United States Department of Defense
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: M-10244
Record Dates: First submitted 2012-11-13; First posted 2012-11-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Traumatic Brain Injury; Brain Concussion
Keywords: DANA; ANAM; Concussion; mild traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-concussed (Active Comparator): Control group; individuals assigned to this group will be either healthy volunteers or individuals sustaining an injury that does not involve concussion. Participants will take both the ANAM and DANA Brief twice at minimum.
  Interventions: Device: DANA Brief; Other: ANAM
- Concussed (Experimental): Individuals who have been diagnosed with a concussion by a clinician. Participants will take both the DANA and ANAM twice at minimum.
  Interventions: Device: DANA Brief; Other: ANAM

INTERVENTIONS:
Device: DANA Brief — The DANA Brief is a newly-developed neurocognitive test administered on a handheld computer that tests simple reaction time, procedural reaction time, code substitution, and spatial processing. The test also includes subtests for depression/distress, PTSD, and insomnia.
Other: ANAM — The ANAM is a currently used test by military health care providers in evaluating cognitive performance after concussion.

SUMMARY:
The Defense Automated Neurobehavioral Assessment (DANA) was recently developed as a durable, portable, and "field-hardened" NeuroCognitive Assessment Tool. The purpose of this study is to compare the sensitivity of the DANA Brief exam with the Automated Neuropsychological Assessment Metrics (ANAM) battery currently used by the military after concussion. The primary hypothesis is that the DANA Brief exam will be more sensitive for detecting continued impaired cognitive performance than the ANAM during recovery after a concussion.

DETAILED DESCRIPTION:
Among active duty military personnel deployed to combat theaters, blast injury is a leading cause of traumatic brain injury (TBI). Service members with TBI can experience notable neurological impairments-e.g., attention disturbances, memory and language deficits, and delayed reaction time. Cognitive performance can still be impaired 2-4 weeks after concussion with no overt physical symptoms. Thus, there is a critical need to have an efficient means to determine the incidence of cognitive deficits in service members exposed to or injured by blasts. To that end, this study plans to evaluate the ANAM and the DANA to determine which neurocognitive test more reliably and accurately detects cognitive impairments during the recovery period from a concussion.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty U.S. military service members
* Clinical diagnosis of concussion/mild traumatic brain injury (mTBI) (as defined by the American Congress of Rehabilitation, 1993, and DoD), made by the treating clinician based on clinical history, examination and/or clinical imaging performed as part of standard of care. This includes subjects with concussion from any mechanism (blast-related, blunt trauma etc.)--for concussed subjects only
* Glasgow Coma Scale (GCS) score of 15 as assessed by the consenting research staff--for concussed subjects only
* Concussive event that occurred within 72 hours of injury (to exclude service members presenting due to lingering effects of a previous injury)--for concussed subjects only
* Willingness to participate in the study, ability to communicate and comply with the study protocol and ability to provide informed consent.

Exclusion Criteria:

* Have a history of other mTBI within 90 days, moderate brain injury within the past 3 years, or any lifetime history of severe brain injury
* History of a documented diagnosis of post traumatic stress disorder (PTSD) or of treatment for PTSD
* Taking psychoactive medications, opioids, or other significant sedating medication
* Individuals with severe psychiatric disorders requiring continuing medication or recent treatment for an alcohol or drug dependency
* Report a pain level of 8 or greater on the 10-point Likert scale of 1 to 10 (e.g., 8, 9 or 10).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evidence of DANA Brief's improved sensitivity compared to ANAM | within 10 days of injury
  Outcome will be confirmed by the ability of the DANA Brief to detect statistically significant differences in cognitive performance between concussed and non-concussed groups even after the ANAM has indicated full recovery

CONTACTS AND LOCATIONS:
Overall Officials: Jack Tsao, MD, DPhil, Principal Investigator — U.S. Navy Bureau of Medicine and Surgery (BUMED)
Locations (1):
- Concussion Restoration Care Center, Camp Leatherneck, Afghanistan